CLINICAL TRIAL: NCT00233792
Title: An Evaluation of the Sirolimus Coated Modified BX VELOCITY Balloon-Expandable Stent in the Treatment of Patients With de Novo or Restenotic Native Coronary Artery Lesions.
Brief Title: FIM-BR - First-in-Man Study (Brazil Part) With Sirolimus-Coated BX VELOCITY Stent
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P99-6301
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2007-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): sirolimus coated Bx VELOCITY stent - fast release
  Interventions: Device: sirolimus coated Bx VELOCITY stent - fast release
- 2 (Other): sirolimus coated Bx VELOCITY stent - slow release
  Interventions: Device: sirolimus coated Bx VELOCITY stent - slow release

INTERVENTIONS:
Device: sirolimus coated Bx VELOCITY stent - fast release
  Arms: 1
Device: sirolimus coated Bx VELOCITY stent - slow release
  Arms: 2

SUMMARY:
This is a single center, non-randomized study. Patients will be treated with the sirolimus coated Bx VELOCITY Balloon-Expandable Stent mounted on the Raptor OTW SDS. Patients will have a repeat angiography at four months and will be followed for twelve months post-procedure.

DETAILED DESCRIPTION:
This is a single center, non-randomized study of the Bx VELOCITY Balloon-Expandable Stent coated with sirolimus (140µg/cm2) and formulated for fast or slow release. The sirolimus coated stent is mounted on the Raptor OTW SDS. Approximately 30 patients with de novo or restenotic native coronary artery lesions <=18mm in length and >=3.0 to >=3.5 mm in diameter by visual estimate who meet all eligibility criteria will be treated with the sirolimus coated Bx VELOCITY stent(s). Patients will be followed for five years post-procedure and will have a repeat angiography at 4 months, 12 months, 24 months, and 48 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS) or a positive ischemia study;
2. Single de novo or restenotic lesion requiring treatment in a major native coronary artery;
3. Target lesion is <=18mm in length (visual estimate);
4. Target lesion is >=3.0mm and <=3.5mm in diameter (visual estimate);
5. Target lesion stenosis is >50% and <100% (visual estimate);

Exclusion Criteria:

1. A Q-wave or non-Q-wave myocardial infarction within the preceding 72 hours unless the CK and CK-MB enzymes are back to normal;
2. Unprotected left main coronary disease with >=50% stenosis;
3. Have an ostial target lesion;
4. Angiographic evidence of thrombus within target lesion;
5. Calcified lesions which cannot be successfully predilated;
6. Ejection fraction <=30%;
7. Target lesion involves bifurcation (either stenosis of both main vessel and major branch or stenosis of just major branch);
8. Totally occluded vessel;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1999-12; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Assessment of in-stent percent diameter stenosis (%DS) measured by quantitative coronary angiography. | post procedure and 6 months

SECONDARY OUTCOMES:
Assessment of lesion morphology by intravascular ultrasound (IVUS). | post procedure and 6 months
Target vessel failure (TVF). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo J Sousa, MD, Principal Investigator — Instituto Dante Pazzanese of Cardiology
Locations (1):
- Instituto Dante Pazzanese of Cardiology, São Paulo, Brazil

REFERENCES:
- [Result] Sousa JE, Costa MA, Sousa AG, Abizaid AC, Seixas AC, Abizaid AS, Feres F, Mattos LA, Falotico R, Jaeger J, Popma JJ, Serruys PW. Two-year angiographic and intravascular ultrasound follow-up after implantation of sirolimus-eluting stents in human coronary arteries. Circulation. 2003 Jan 28;107(3):381-3. doi: 10.1161/01.cir.0000051720.59095.6d. PMID 12551858
- [Result] Sousa JE, Costa MA, Abizaid A, Feres F, Seixas AC, Tanajura LF, Mattos LA, Falotico R, Jaeger J, Popma JJ, Serruys PW, Sousa AG. Four-year angiographic and intravascular ultrasound follow-up of patients treated with sirolimus-eluting stents. Circulation. 2005 May 10;111(18):2326-9. doi: 10.1161/01.CIR.0000164271.01172.1A. Epub 2005 Apr 25. PMID 15851603
- [Result] Aoki J, Abizaid AC, Serruys PW, Ong AT, Boersma E, Sousa JE, Bruining N. Evaluation of four-year coronary artery response after sirolimus-eluting stent implantation using serial quantitative intravascular ultrasound and computer-assisted grayscale value analysis for plaque composition in event-free patients. J Am Coll Cardiol. 2005 Nov 1;46(9):1670-6. doi: 10.1016/j.jacc.2005.06.076. Epub 2005 Oct 10. PMID 16256867
- [Result] Sousa JE, Costa MA, Abizaid A, Abizaid AS, Feres F, Pinto IM, Seixas AC, Staico R, Mattos LA, Sousa AG, Falotico R, Jaeger J, Popma JJ, Serruys PW. Lack of neointimal proliferation after implantation of sirolimus-coated stents in human coronary arteries: a quantitative coronary angiography and three-dimensional intravascular ultrasound study. Circulation. 2001 Jan 16;103(2):192-5. doi: 10.1161/01.cir.103.2.192. PMID 11208675